CLINICAL TRIAL: NCT06519370
Title: A Phase 3, Open-label, Randomised Study of FDA018-ADC Versus Investigator's Choice of Chemotherapy in Patients Who Recurred During or After Taxane Therapy in Locally Advanced or Metastatic Triple-negative Breast Cancer
Brief Title: FDA018-ADC vs Investigator's Choice Chemotherapy to Treat Locally Advanced, Recurrent or Metastatic Triple-negative Breast Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Fudan-Zhangjiang Bio-Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F0024-301
Record Dates: First submitted 2024-07-18; First posted 2024-07-25 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — eribulin; Capecitabine; Gemcitabine; Vinorelbine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FDA018-ADC (Experimental): Subjects will receive FDA018-ADC 10 mg/kg of body weight via intravenous(IV) infusion on Day1 and 8 of a 21-day cycle in follow-up period until disease progression, unacceptable toxicity or death.
  Interventions: Drug: FDA018-ADC
- Investigator's Choice of Chemotherapy (ICC) (Active Comparator): Participants will receive ICC (ie, eribulin, capecitabine, gemcitabine, or vinorelbine), administered as a single-agent regimen that is selected by the investigator before participant randomization. Participants will continue treatment until disease progression, unacceptable toxicity or death.
  Interventions: Drug: Eribulin; Drug: Capecitabine; Drug: Gemcitabine; Drug: Vinorelbine

INTERVENTIONS:
Drug: FDA018-ADC — Subjects will receive FDA018-ADC 10 mg/kg of body weight via intravenous(IV) infusion on Day1 and 8 of a 21-day cycle in follow-up period until disease progression, unacceptable toxicity or death.
  Other Names: FDA018-Antibody-drug Conjugate
  Arms: FDA018-ADC
Drug: Eribulin — 1.4mg/m^2, IV (in the vein) on day 1 and Day 8 of each 21 day cycle
  Other Names: Halaven
  Arms: Investigator's Choice of Chemotherapy (ICC)
Drug: Capecitabine — 1000 to 1250 mg/m^2 will be administered in a 21-day cycle, with capecitabine administered orally twice daily for 2 weeks followed by 1-week rest
  Other Names: Xeloda
  Arms: Investigator's Choice of Chemotherapy (ICC)
Drug: Gemcitabine — 800 to 1200 mg/m^2 will be administered IV on day 1 and Day 8 of each 21 day cycle
  Other Names: Gemzar
  Arms: Investigator's Choice of Chemotherapy (ICC)
Drug: Vinorelbine — 25 mg/m^2, IV (in the vein) on day 1 and Day 8 of each 21 day cycle
  Other Names: Navelbine
  Arms: Investigator's Choice of Chemotherapy (ICC)

SUMMARY:
This is a Phase III, randomized, open-label, 2-arm, multicentre, international study assessing the efficacy and safety of FDA018-ADC compared with Investigator's Choice Chemotherapy(ICC) in participants with locally recurrent inoperable or metastatic Triple-negative Breast Cancer(TNBC) who are resistant to, or recurring during or after taxane therapy.

DETAILED DESCRIPTION:
The primary objectives of the study are to demonstrate the superiority of FDA018-ADC relative to ICC by assessment of PFS per Blinded Independent Central Review(BICR) and OS in participants with locally recurrent inoperable or metastatic TNBC who are resistant to, or recurring during or after taxane therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients capable to give written informed consent;
2. Histologically or cytologically confirmed TNBC based on the most recent analyzed biopsy or other pathology specimen. Triple negative is defined as <1% expression for estrogen receptor (ER) and progesterone receptor (PR) and negative for human epidermal growth factor receptor 2 (HER2) by in-situ hybridization;
3. Prior exposure to a taxane in localized or advanced/metastatic setting, and recurred during or after treatment;
4. Eligible for one of the chemotherapy options listed as ICC (eribulin, capecitabine, gemcitabine, or vinorelbine) as per investigator assessment;
5. Have measurable lesions defined in RECIST v.1.1, those with only skin or bone lesions cannot be included;
6. Expected survival≥3 months;
7. Eastern Cancer Cooperative Group (ECOG) performance status 0-1;
8. Adequate bone marrow, hepatic, and renal function;
9. All acute toxicity of previous anti-tumor treatment or surgery is relieved to baseline severity or NCI CTCAE version 5.0≤1;
10. Subjects could provide tumor tissues or tissue specimens;
11. Patients of child bearing potential must agree to take contraception during the study and for 6 months after the last day of treatment.

Exclusion Criteria:

1. Patients with other malignancies, except cured basal or squamous cell skin cancer or in situ cancer of cervix; and patients with other malignancies must have a tumor-free period of at least 5 years;
2. Have central nervous system metastasis with clinical symptoms;
3. Have history of clinical significant active chronic obstructive pulmonary disease, or other moderate-to-severe chronic respiratory illness present within 6 months prior to the first dose;
4. Suffering from active chronic inflammatory bowel disease (ulcerative colitis, Crohn disease), and history of intestinal obstruction, or Gl perforation;
5. Patients with Gilbert's disease or heterozygous for the UGT1A1*28 allele;
6. Participants known to be human immunodeficiency (HIV) positive, hepatitis B positive, or hepatitis C positive;
7. Patients who have received prior TROP-2-targeted therapy;
8. Patients who have received prior topoisomerase I inhibitor contained therapy;
9. Received other anti-tumor treatments (including chemotherapy, radiotherapy, targeted therapy, immunotherapy, experimental treatment and so on) within 4 weeks prior to the first dose;
10. Patients who have received live vaccines within 4 weeks prior to the first dose;
11. Patients who had undergone major surgery or severe trauma within 4 weeks prior to the first dose;
12. Patients who had undergone systemic high-dose steroids within 2 weeks prior to the first dose;
13. Patients have history of psychotropic drug abuse, alcohol or drug abuse;
14. Women who are pregnant or lactating;
15. Other circumstances that is deemed not appropriate for the study by investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2024-08-09 (Actual); Primary Completion 2026-08-18 (Estimated); Study Completion 2027-06-20 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | up to 24 months
  PFS is defined as time from randomisation until progression per RECIST 1.1 as assessed by BICR, or death due to any cause
Overall Survival (OS) | up to 24 months
  OS is defined as the time from randomisation until the date of death due to any cause.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) by Investigator assessment | up to 24 months
  PFS is defined as time from randomisation until progression per RECIST 1.1 as assessed by the investigator, or death due to any cause
Objective Response Rate (ORR) | up to 24 months
  ORR is defined as the proportion of participants who have a confirmed CR or PR, as determined by BICR/investigator assessment, per RECIST 1.1.
Duration of Response Duration of Response (DoR) | up to 24 months
  DoR is defined as the time from the date of first documented confirmed response until date of documented progression per RECIST 1.1, as assessed by BICR/investigator assessment or death due to any cause.
Disease Control Rate (DCR) | up to 24 months
  DCR is defined as the proportion of patients who have achieved complete response，partial response and stable disease assessed by BICR/investigator according to RECIST v 1.1
Incidence of Treatment-Emergent Adverse Events | up to 24 months
  Incidence and severity of AEs and SAEs (graded by CTCAE version 5.0).
Immunogenicity of FDA018-ADC | up to 24 months
  Presence of ADAs for FDA018-ADC

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhang, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No